CLINICAL TRIAL: NCT02406365
Title: Development and Application of a Diagnostic Imaging Aid for One-visit Management of Cervical Lesions in Low-resource Settings
Brief Title: Diagnostic Imaging Aid for Management of Cervical Lesions
Acronym: FFC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brookdale University Hospital Medical Center (Other)
Responsible Party: Principal Investigator, Michele Follen, Chair of Department of Obstetrics and Gynecology, Brookdale University Hospital Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-36
Record Dates: First submitted 2015-03-17; First posted 2015-04-02 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Cervical Cancer; Cervical Intraepithelial Neoplasias; Digital Colposcopy; Precancerous Cervical Lesions
MeSH Terms: conditions — Uterine Cervical Neoplasms

ARMS (1):
- Standard of care plus imaging with research devices (Experimental): Eligible patients who consent to participate in the research study will receive their standard of care colposcopy or treatment with the Loop Electrosurgical Excision Procedure (LEEP). Additionally, cervical images will be taken using the diagnostic imaging aid. The cervical images will be compared to the histopathology from the biopsies taken as part of the patients' standard of care for colposcopy. If the patient is presenting for the LEEP procedure, then she will be asked if one or two biopsies can be obtained prior to the procedure but after anesthesia has been administered.
  The imaging device is not being used to make a diagnosis, but rather to develop an algorithm to make more efficacious and timely diagnoses of cervical neoplasias in the future.
  Interventions: Device: Diagnostic imaging aid for one-visit management of cervical lesions

INTERVENTIONS:
Device: Diagnostic imaging aid for one-visit management of cervical lesions

SUMMARY:
A handheld digital colposcope which utilizes flurorescent light is being tested for the rapid detection and management of cervical lesions. The handheld research device captures cervical images which with the fluorescent light show the regions of cervical tissue that autofluoresce. The investigators will study the relationship between the level of fluorescence and the samples of tissue (biopsies) obtained from the patient as part of her routine care. The investigators will also compare the efficacy of the hand held device with the data being collected from the other research devices being tested by the team, i.e. the multispectral digital colposcopes.

ELIGIBILITY:
Inclusion Criteria:

* Women who are at least 18 years old
* Women who are not pregnant as confirmed by a urine test
* Women who are not breastfeeding
* Women who understand the study procedures and can provide written informed consent

Exclusion Criteria:

* Women who do not meet the inclusion criteria
* Women who have had a hysterectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 618 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Detection of precancerous cervical lesions or cervical cancer | At point of care for colposcopy or treatment with LEEP (5 minutes).
  Eligible patients who are referred to the colposcopy clinic for a diagnosis following an abnormal Pap smear will be asked to participate in the study. All participating women will receive their standard of care colposcopy as usual. In addition to their routine care, the handheld imaging research device will also be used to capture cervical images. The images will be analyzed and compared to the biopsies obtained. The imaging device will not be used to make a diagnosis. As part of the research study, one or two additional biopsies will be obtained if the patient agrees. These additional biopsies will serve as the control tissue, since they will be taken from tissue that appears normal through the colposcope.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Follen, PhD, Principal Investigator — Brookdale University Hospital and Medical Center
Locations (1):
- Brookdale University Hospital and Medical Center, Brooklyn, New York, United States